CLINICAL TRIAL: NCT06485817
Title: How Distress Alters Opioid Drug Effects and Abuse Liability
Brief Title: How Stress Alters Opioid Drug Effects
Acronym: OPIOIDREWARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: Oslo University Hospital (Other); Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Marie Eikemo, Co-Principal Investigator, University of Oslo
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Basic Science
Other Study IDs: 802885; https://osf.io/bcxv8 (Other: OSF)
Record Dates: First submitted 2024-06-07; First posted 2024-07-03 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Motivation; Drug Effect; Stress Reaction; Misuse, Opioid
MeSH Terms: conditions — Fractures, Stress; Opioid-Related Disorders | interventions — Oxycodone; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Cross-over 2*2 design Drug (i.v. oxycodone/placebo) State induction (stress/control)
Who Masked: Participant, Care Provider, Investigator
Masking Description: Experimenters, care providers (nurses/physicians) and participants were blinded to both the stress induction condition and the drug in all sessions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo_Control (Placebo Comparator): Control state induction:
  Participants answer simple questions about their color or music preferences in a hybrid (zoom-lab) session with a friendly experimenter (The Repeatable Social Stress Test (ReSST) control conditions).
  Drug administration:
  A sampling dose of intravenous (i.v.) saline administered over 15 seconds through a venous catheter after the state induction. 45 minutes later participants receive the second dose of saline (0-100% of the initial sampling dose) determined by a behavioral self-administration task.
  Interventions: Drug: Placebo; Behavioral: Control State Induction
- Oxycodone_Control (Active Comparator): Control state induction:
  Participants answer simple questions about their color or music preferences in a hybrid (zoom-lab) session with a friendly experimenter. (The Repeatable Social Stress Test (ReSST) control conditions).
  Drug administration:
  A sampling dose of i.v. oxycodone administered over 15 seconds through a venous catheter after the state induction. 45 minutes later participants receive the second dose of oxycodone (0-100% of the initial sampling dose) determined by a behavioral self-administration task.
  Interventions: Drug: Oxycodone; Behavioral: Control State Induction
- Placebo_Stress (Active Comparator): State induction: Stress The Repeatable Social Stress Test (ReSST) was used to induce psychosocial stress (mock job talk in stress session 1 and singing task in stress session 2).
  Drug administration:
  A sampling dose of i.v. saline administered over 15 seconds through a venous catheter after the state induction. 45 minutes later participants receive the second dose of saline (0-100% of the initial sampling dose) determined by a behavioral self-administration task.
  Interventions: Drug: Placebo; Behavioral: Stress State Induction
- Oxycodone_Stress (Experimental): State induction: Stress ReSST was used to induce psychosocial stress (mock job talk in stress session 1 and singing task in stress session 2).
  Drug administration:
  A sampling dose of i.v. oxycodone administered over 15 seconds through a venous catheter after the state induction. 45 minutes later participants receive the second dose of oxycodone (0-100% of the initial sampling dose) determined by a behavioral self-administration task.
  Interventions: Drug: Oxycodone; Behavioral: Stress State Induction

INTERVENTIONS:
Drug: Oxycodone — 3.1mg oxycodone/70 kg body weight was administered as the main drug intervention.
  Based on body weight, the study nurse/anesthetist adjusted the (unknown) content in two syringes by removing enough fluid to reach a volume that would result in a dose equivalent of 3.1mg/70kg (0,043 mg/ml pr kg) should the syringes contain oxycodone.
  The first dose was administered 5 minutes after the state induction task. The second dose was adjusted according to the performance on the self-administration task (but maximum 100% of the first dose) and administered 45 later.
  Arms: Oxycodone_Control; Oxycodone_Stress
Drug: Placebo — Pure saline was administered as the placebo condition.
  Based on body weight, the study nurse/anesthetist adjusted the (unknown) content in two syringes by removing enough fluid to reach a volume that would result in a dose equivalent of 3.1mg/70kg (0,043 mg/ml pr kg) should the syringes contain oxycodone.
  The first dose was administered 5 minutes after the state induction task. The second dose was adjusted according to the performance on the self-administration task (but maximum 100% of the first dose) and administered 45 later.
  Other Names: Saline
  Arms: Placebo_Control; Placebo_Stress
Behavioral: Stress State Induction — ReSST is an in-house hybrid online-lab implementation of two stress induction paradigms based on the Trier Social stress test (TSST) and Iowa Social Singing Stress Test (I-SSST).
  The set-up was tailored to allow repeated stress induction without diminishing effects that allowed for an online experiment panel. Stress and control state inductions were administered every-other session. The singing version of the stress test was always administered last as it was deemed more stressful during piloting.
  Other Names: ReSST (Repeatable Social Stress Test): Stress
  Arms: Oxycodone_Stress; Placebo_Stress
Behavioral: Control State Induction — Two different control tasks matched to the stress conditions on key parameters outlined in the protocol.
  Other Names: ReSST (Repeatable Social Stress Test): Control
  Arms: Oxycodone_Control; Placebo_Control

SUMMARY:
The main objective of the study is to test the hypothesis that opioid drug effects vary as a function of pre-drug affective state. Specifically, it is hypothesized that social stress induction enhances opioid drug wanting compared a non-stress control condition.

DETAILED DESCRIPTION:
Healthy participants complete four experiment sessions in a placebo-controlled, double-blind, randomized repeated-measures psychopharmacological study. Participants completed four combinations of pre-drug state induction (social stress or no-stress) and drug (intravenous oxycodone or saline).

Temporary and reversible social stress is induced using the Repeatable Social Stress Test (ReSST) which enables repeated administrations of stress-inductions. Across four sessions participants experience two carefully tailored tasks to provoke the experience of social evaluative threat and two non-stressful control tasks.

After each state inductions, participants receive an injection of opioid drug or saline. After a drug absorption phase and viewing of a state reinstatement video designed to evoke a mild form of social evaluative threat participants perform a drug-self-administration test to determine the potency of a second dose.

Self-reported affect, mental and physiological state and drug effects are assessed throughout the session.

ELIGIBILITY:
Inclusion Criteria:

* Mentally and physically healthy
* Body mass index (BMI) in the healthy range (18.5 < BMI < 30)
* Normal or corrected vision
* Had received an opioid drug at least once in their lifetime (to ensure no severe adverse or allergic reactions).

Exclusion Criteria:

* Any significant physical health problem (e.g., heart, lung, kidney, liver, and other conditions)
* Current or past substance use problems
* Current mental health problems
* Past mental health problems beyond mild episodic anxiety or depression
* Social anxiety or fear of public speaking
* Past or current chronic pain
* Pregnancy or breastfeeding
* Recent use of any contraindicating medications
* Prior difficulty in providing blood samples.

All exclusion criteria required a 'yes' or 'no' response from participants. Participants were also asked to report any illnesses or medical conditions that were not covered by the questions in the clinical interview. Mental health and substance use were assessed during the clinical interview using the Mini-International Neuropsychiatric Interview (MINI). The interview required binary responses to questions regarding a wide range of psychological symptoms relevant for DSM-IV (Diagnostic and Statistical Manual of Mental Disorders) and ICD-10 (International Classification of Diseases) psychiatric disorders. Interviewers then used the pre-defined cut offs relevant to the severity of symptoms for each psychiatric disorder to assist the clinical judgement.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2022-04-28 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Amount of oxycodone self-administered in the behavioral drug wanting task relative to the first sampling dose (0-125%). | Single measure: final task result ~22 minutes after sampling dose
  The number corresponds to the achieved cursor placement on a vertical electronic scale indicated desired effect intensity from second dose relative to the first (sampling) dose. Cursor placement depends on the amount of effort exerted (keyboard presses) and the task difficulty adapted to performance. The task ended abruptly after 2 minutes.
Self-report of oxycodone wanting relative to the first sampling dose (0-125 %) | Single measure: ~20 minutes after sampling dose
  Self-reported target effect intensity was indicated on a vertical scale at the onset of the behavioral drug wanting task before the effortful part of the task.
  Anchors visible to to participants were: "no effect/drug", "half the effect", "same effect", "a little stronger effect than the first drug dose". Numerically the scale anchors were 0-125 (VAS) where 100 corresponded to the "same effect".
Self-reported drug wanting from "drug effects questionnaire". | From the drug administration until the start of the self-administration task (~15 minutes)
  Drug effects questionnaire (DEQ) take again item indicated on a 0-100 electronic Visual analogue scale (VAS) at two survey timepoints after the drug administration. Anchors were 'neutral' and 'very much'. Average rating was used.

SECONDARY OUTCOMES:
Stress response 1: increase in self-reported stress to the primary stress induction and subsequent stress reinstatement (as compared to control tasks). | From the measure before state induction until the end of the state induction (~20 minutes).
  Change in ratings on the item "feeling stressed" measured on a 0-100 Visual Analogue Scale (VAS) The following items were collected to assess stress effects: anxious, self-conscious, embarrassed, vulnerable, happy, relaxed, irritable, confident, shaky, distressed, flushed face, heart palpitations, stomach discomfort, dizzy (to stress on a 0-100 VAS) and report this in the supplementary materials.
Stress response 2: increase in physiological stress measured by heart rate (beats per minute: BMP) induced by the primary stress induction. | Data from 20 minutes before to 20 minutes after the middle of the stress induction were used to estimate the heart rate increase
  Heart rate change during the state induction compared to the time period before state induction.
Stress response 3: change in endocrine stress response measured by cortisol induced by the primary stress induction. | Throughout the experiment session (~3 hours, 6 samples)
  Estimates of plasma cortisol levels changes from the baseline (2 blood samples) to the samples after the state induction (4 blood samples).
Changes in positive and negative affect after the state manipulations (induction and reinstatement) and drug administrations | From immediately before to immediately after the state induction (~20 minutes)
  Select items from the PANAS based on pilot data. Baseline measures are collected several times before the state induction. Items were rated on a 0-100 Visual Analogue Scale (VAS).
  Negative affect (mood) items = "distressed", "anxious", "vulnerable", "irritable" Positive affect (mood) items = "good", "happy", "confident", "safe", "relaxed"
  Composite ratings from all measures collected throughout each session (k=11 measures) will be reported as descriptive information.
Drug effects questionnaire (DEQ) | From the drug administration until the start of the self-administration task (~15 minutes)
  Drug effect, liking and disliking was measured using items from the Drug Effects Questionnaire (DEQ; 'Feel effect', 'Like effect', 'Dislike effect') measured on an electronic 0-100 VAS, anchors 'neutral' and 'very much'.
Side effects | From the drug administration until the start of the self-administration task (~15 minutes)
  To assess the overall drug- and side effects, the following items were collected on a 0-100 electronic VAS: feeling high, blunted and dizzy.
  Additional items will be explored and reported where relevant and in the supplementary materials (feeling good, euphoric, indifferent, safe, dry mouth, nauseous, "not like myself").

CONTACTS AND LOCATIONS:
Overall Officials: Siri Leknes, PhD, Principal Investigator — University of Oslo; Marie Eikemo, PhD, Principal Investigator — University of Oslo
Locations (1):
- University of Oslo, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
Anonymized information (non sensitive) will be shared on the Open Science Framework (OSF) at the time of publication.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: The data will be released with the publication. The code, protocol, and supplementary materials have been released in the project repository.
Access Criteria: none. For conditional access to health/sensitive data following publication contact the corresponding author (marie.eikemo@psykologi.uio.no) A data use agreement may also be required.
URL: https://osf.io/3jvw8/

REFERENCES:
- See also: Time locked preregistration prior to data collection — https://osf.io/bcxv8/
- Available data/document: Analytic Code — https://osf.io/3jvw8/ — Project directory where study relevant documentation can be found and data will be uploaded.